CLINICAL TRIAL: NCT06366399
Title: Timing (AM v PM) of Acute Resistance Exercise on Glycemic Control in Older Adults: The Acute T-Rex Study
Brief Title: The Acute T-Rex (Timing of Resistance Exercise) Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 00156659
Record Dates: First submitted 2024-01-31; First posted 2024-04-15 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Diabetes Mellitus, Type 2; Insulin Resistance; Glucose Intolerance; Sleep Disturbance; Overweight or Obesity; Insulin Sensitivity
Keywords: Resistance Exercise; Strength-training; Sleep; Circadian Rhythm
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance; Glucose Intolerance; Parasomnias; Overweight; Obesity | interventions — Exercise; Resistance Training

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AM Resistance Exercise (Experimental): Resistance Exercise intervention taking place in the AM
  Interventions: Behavioral: Resistance Exercise Timing
- PM Resistance Exercise (Experimental): Resistance Exercise intervention taking place in the PM
  Interventions: Behavioral: Resistance Exercise Timing

INTERVENTIONS:
Behavioral: Resistance Exercise Timing — 1 resistance exercise session consisting of 3 sets, 10 repetitions per set, on 12 different exercises
  Other Names: Exercise; Strength-Training; Weightlifting

SUMMARY:
The primary aim of this study is to evaluate if a single bout of AM vs PM resistance exercise has different effects on insulin sensitivity and sleep. A randomized cross-over trial be used to compare resistance exercise at two different times of the day. Each condition will take place in a laboratory setting. Each condition will consist of exercise, overnight sleep, and oral glucose tolerance tests the following day. The AM exercise will occur ~1.5 hours after habitual wake, and PM exercise will occur ~11 hours after habitual wake. After a 2-6 week washout, participants will complete the other condition. The hypothesis is that PM exercise will be more beneficial than AM exercise in improving insulin sensitivity. This study could identify if there is a better time of day to perform resistance exercise to decrease risk of developing Type 2 Diabetes Mellitus.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, all ethnicities, aged 50-74 years
* BMI ≥25 kg/m² and <45 kg/m²
* Weight stable (less than 5% change in the past 6 months)
* Generally healthy individuals
* Not meeting recommended activity guidelines for aerobic or resistance exercise

Exclusion Criteria:

* Uncontrolled cardiovascular, metabolic, renal, or pulmonary disease
* Cancer treatment in the past 5 years
* Untreated thyroid disease or other medical conditions affecting weight or energy metabolism
* Current use of weight loss medication or other medications likely to impact energy balance
* Bariatric surgery or extensive bowel resection in the past 2 years
* Current or recent history (past 2 years) of eating disorder
* Diagnosis of insomnia, sleep apnea, or other sleep and circadian disorders
* Non-English speaking
* HbA1c >6.5%

Ages: 50 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-11-15 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Insulin sensitivity | 1 day
  Insulin sensitivity will be calculated using the Matsuda Insulin Sensitivity Index

SECONDARY OUTCOMES:
Sleep Duration | 1 day
  Sum of time spent in stage 1, stage 2, stage 3 and rapid eye movement stage (REM) as assessed via polysomnography.

OTHER OUTCOMES:
Sleep Staging | 1 day
  Time spent in stage 1, stage 2, stage 3 and REM sleep assessed by polysomnography.
Sleep Quality | 1 day
  As assessed via Pittsburg Sleep Quality Index Questionnaire (scale:0-21, higher scores=worse outcome) and polysomnography
Sleep Efficiency | 1 day
  Ratio of time in bed vs time asleep
Muscular Strength | 1 day
  Muscular strength as assessed via 10 repetition maximum test
Perceived Hunger | 1 day
  Visual Analog Scales (scale: 0-100)
Perceived Fullness | 1 day
  Visual Analog Scales (scale: 0-100)
Perceived Prospective Food Consumption | 1 day
  Visual Analog Scales (scale: 0-100)
Glucose Area Under Curve | 1 day
  Mathematical calculation using fasting, 10,20,30,60,90,120 min blood glucose
Insulin Area Under Curve | 1 day
  Mathematical calculation using fasting, 10,20,30,60,90,120 min blood insulin

CONTACTS AND LOCATIONS:
Locations (1):
- University of Utah HPER E Buildling, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No